CLINICAL TRIAL: NCT01152242
Title: A Two-Part Clinical Trial to Assess Pharmacodynamic and Pharmacokinetic Variability of a Basal Insulin
Brief Title: Pharmacodynamic and Pharmacokinetic Variability of a Basal Insulin (0000-168)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0000-168; 2010_541 (Other: Merck)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: Insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Active Comparator): Part I of the trial
  Interventions: Drug: Isoglycemic Clamp; Drug: Comparator: insulin glargine
- Part 2 (Active Comparator): Part II of the trial
  Interventions: Drug: Isoglycemic Clamp; Drug: Comparator: insulin glargine

INTERVENTIONS:
Drug: Isoglycemic Clamp — Isoglycemic Clamp, a procedure that includes IV infusion of short-acting Insulin (Part I) and glucose (Part I and 2)
Drug: Comparator: insulin glargine — Insulin glargine at 0.4 U/kg
  Other Names: LANTUS

SUMMARY:
The purpose of this study is to evaluate whether the within-subject variation in duration of action and time-action profile of glargine measured by isoglycemic clamp will be below prespecified levels.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Patient is a male between 18 to 45 years of age (inclusive) at the prestudy (screening) visit
* Patient has a clinical diagnosis of type 1 diabetes
* Patient must have been treated with insulin since diagnosis and be on a stable dose of insulin
* Patient has a Body Mass Index (BMI) of <=27 kg/m2 and >18 kg/m2
* Patient has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Part 2:

* Subject is a male between 18 to 45 years of age at the prestudy (screening) visit
* Subject has a Body Mass Index (BMI) of <=25 kg/m^2
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months

Exclusion Criteria:

Part 1:

* Patient has a history of stroke, chronic seizures, or major neurological disorder
* Patient has currently active and untreated clinically significant endocrine, cardiovascular, hematological, hepatic, renal, respiratory, or genitourinary abnormalities or diseases
* Patient has a history of hypertension requiring treatment
* Patient has a history of neoplastic disease within the past 5 years
* Patient is currently being treated with, or has a history of treatment with any oral antihyperglycemic agent
* Patient has a history of significant multiple and/or severe allergies

Part 2:

* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of hypertension requiring treatment
* Subject has a history of neoplastic disease within the past 5 years
* Subject has history of diabetes (Type 1, Type 2 or steroid-induced) or family history of diabetes mellitus
* Subject has a history of hypersensitivity to glargine or any of its inactive ingredients

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Part I: The within-subject standard deviation in duration of action of glargine (the difference between onset of action and end of action) | Baseline and 30 hours
Part II: The within-subject coefficient of variation in time-action profile of glargine for AUC-GIR (AUC of glucose infusion rate), GIRmax (maximum level of glucose infusion rate), over the duration of action of glargine | Baseline and 30 hours

SECONDARY OUTCOMES:
Part I: The within-subject coefficient of variation in time-action profile of glargine for AUC-GIR and GIRmax over the duration of action of glargine | Baseline and 30 hours
Part II: The within-subject standard deviation in duration of action of glargine (the difference between onset of action and end of action) | Baseline and 30 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC